CLINICAL TRIAL: NCT06309524
Title: Valutazione Del Rimodellamento Delle Camere Destre Dopo Trattamento Transcatetere Edge-to-edge Dell'Insufficienza Tricuspidale Severa
Brief Title: Assessing the Right Heart Remodeling After Transcatheter Tricuspid Edge-to-edge Repair
Acronym: HERITAGE
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C332
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Tricuspid transcatheter edge-to-edge repair — Transcatheter tricuspid leaflets approximation

SUMMARY:
In the recent years, secondary tricuspid regurgitation (STR) has gained interest due to its high prevalence and impact on outcomes. Transcatheter tricuspid valve replacement or repair represents novel and less invasive alternatives to surgery and has shown early promising results. Treatment options mimic surgical techniques such as leaflet approximation, direct annuloplasty, and heterotopic caval valve implantation, as well as not yet commercially available transcatheter TV replacement systems using orthotopic valve implantation. (5) Among leaflet approximation techniques, the Tricuspid transcatheter edge-to-edge repair (T-TEER) using the TriClip™ (Abbott Vascular, Santa Clara, CA, USA) or leaflet approximation with the PASCAL systems (Edwards Lifesciences, Irvine, CA, USA) are approved in Europe for minimally invasive TV repair.The purposes of the present study are: i. to use 3DE and CCT to evaluate the effect of T-TEER on the geometry and function of the right heart chambers in patients with STR; ii. to identify the predictors of procedural success potentially related to features of both right chambers geometry and TR jet; iii. to compare the accuracy of 3DE assessment of the right ventricle, the right atrium, and the tricuspid annulus, with the same parameters obtained by CCT, in the setting of T-TEER; and iv. to assess patients' outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Severe STR, amenable to percutaneous treatment with T-TEER
* Acceptance to be part of this study by signing the informed consent
* Good enough acoustic window and ability to cooperate in order to obtain 3D echo data sets of cardiac structures with a minimum temporal resolution of 20 fps
* Availability for clinical, CCT and, echocardiography follow-up visits

Exclusion Criteria:

* Pregnancy
* Severe chronic kidney disease (GFR <30 mL/min)
* Hypersensitivity reactions to contrast media
* Cardiovascular implantable electronic device-related (CIED) tricuspid regurgitation.
* Bad acoustic window with inadequate echocardiographic images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic tricuspid regurgitation that fulfill Guidelines criteria for transcatheter tricuspid valve repair
Sampling Method: Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Inverse remodeling of right heart chambers | At baseline and at 6 months after intervention
  Change in inverse remodeling of right heart chambers at 6 months after intervention
Heart failure hospitalization | During 6 months after intervention
  Incidence of heart failure hospitalization during 6 months after intervention
Death | During 6 months after intervention
  Incidence of death during 6 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Lombardy, Italy